**Study Title:** Expressive Helping for Chinese-Speaking Cancer Patients and Survivors

NCT Number: NCT05456100

**Document Date:** 01/24/2025



Applied Psychology 246 Greene St. 8th Floor New York, NY 10003 P: 212-998-4808 Will.tsai@nyu.edu

# Consent to Participate in Research Form for IRB-FY2020-4194

You are invited to take part in a research study to learn about your experiences as a Chinese cancer survivor. This research is being done because many people report physical symptoms and emotional distress even after completing cancer treatment. Past research shows that certain ways of writing can reduce these kinds of symptoms. The purpose of this study is to compare the effects of three different types of writing to see how each one affects physical symptoms and emotional distress. This study will be conducted by William Tsai, Ph.D., from the Department of Applied Psychology in Steinhardt School of Culture, Education, and Human Development, New York University.

#### Who can participate?

You can participate in this study if you match ALL of the following criteria:

- Of Chinese descent
- Living in the United States
- 18 years to 80 years old
- Can read and write in Chinese
- Completed cancer treatment within last five years or have completed primary treatment but still on medication for managing cancer-related symptoms.

### What will happen if I take part in this research study and how long will it take?

- 1. You will complete an online survey that takes approximately 45 minutes. This survey will ask about a variety of topics including your health and life experiences.
- 2. You will complete four 20-minute online writing sessions designed for us to understand your experience as a cancer survivor. These writing sessions are spread out over four weeks (one per week for a total of four weeks).
- 3. You will be asked to complete three follow-up online surveys at one, three, and six months after you have completed the writing sessions. These surveys are similar to the questions you have answered at the beginning of the study. Each survey will take about 30 minutes to finish.
- 4. After you finish the six-month follow-up survey, you may be invited to complete a 30-minute phone interview to provide us with your feedback about the study and for us to better understand your cancer experience.

Before you start writing, you will be "randomized" into one of three writing groups. All groups will involve writing about your cancer experiences. However, the groups will receive different writing instructions. Randomization means that you are put into a group by chance. It is like flipping a coin. A computer is used to assign you to a group. Neither you nor the researchers choose what group you will be in. You will have an equal chance of being placed in either of the three groups. The researcher you speak with will not know what group you are in.

In total, participation in this study will involve about 4 hours of your time: 45 minutes to complete the survey #1, 80 minutes total to complete the 4 writing sessions, 30 minutes to complete survey #2 (sent one month after writing), 30 minutes to complete survey #3 (sent two months after survey #2), and 30 minutes to complete survey #4 (sent three months after survey #3). A small number of participants will be invited to complete a 30 minutes phone interview.

#### Are there any potential benefits if I participate?

You may not directly benefit from participating in this study. However, people have often reported that writing about their cancer experiences is a positive experience. Even if you do not benefit personally, your

NYU IRB-FY2020-4194 Approved on 1-24-2025 Expires on 1-24-2026

**Applied Psychology** 246 Greene St 8th Floor New York, NY 10003 P: 212-998-4808 Will.tsai@nyu.edu

participation will better help the researchers understand the experiences of Chinese cancer survivors as few studies are available for this population.

#### Are there any potential risks if I participate?

It is possible that writing about your cancer experiences and answering survey items and interview questions about your well-being may bring up negative emotions, but this is a rare risk. To minimize this risk, please remember that you can skip any questions you don't want to answer and that you may withdraw from the study at any time without any penalty.

# What happens if I withdraw from the study?

If you withdraw from the study, then the researchers will stop sending you the writing instructions and you will no longer be able to participate in the writing sessions.

The researchers may withdraw you from the study if the participant does not complete the writing sessions as requested. If the researchers withdraw you from the study, then they will stop sending you the writing instructions and you will no longer be able to participate in the writing sessions.

### What other options are there?

The alternative to participation is not to participate in this research.

### Will I receive any payment if I participate in this study?

In total, you can receive up to \$120 in prepaid Visa Debit cards. You will receive \$50 prepaid Visa Debit card for completing the first survey and four 20-minute writing sessions. You will receive a \$20 prepaid Visa Debit card for completing the 1-month follow-up survey, another \$20 prepaid Visa Debit card for completing the 3month follow-up survey, and another \$20 prepaid Visa Debit card for completing the six-month follow-up survey. Lastly, you will receive \$10 prepaid Visa Debit card for completing the 30-minute interview.

#### Will information about me and my participation be kept confidential?

Confidentiality of your research records will be strictly maintained. You will not be identified in any reports on this study and your responses to the surveys will only be identified by a unique number that cannot be linked back to your personal information. Your research records will be stored in a locked file cabinet and in a password-protected database on a secure research server. Only the research team will know that you participated in this study and have access to the research data. With your permission, excerpts from your writing sessions may be shared with others, but your personal information (e.g., name) and survey will not be shared with others. This research is covered by a Certificate of Confidentiality from the National Institutes of Health. Researchers with this Certificate will not disclose or use information that may identify you in any federal, state, or local civil, criminal, administrative, legislative, or other action, suit, or proceeding, even if there is a court subpoena.

#### Exceptions include:

A federal, state, or local law requires disclosure.

Your explicit approval for the researchers to release your name and or personally identifiable information.

A description of this clinical trial will be available on http://www.ClinicalTrials.gov, as required by U.S. Law. This Web site will not include information that can identify you. At most, the Website will include a summary of the results. You can search this Website at any time. Information not containing identifiers may be used in future research, shared with other researchers, or placed in a data repository without your additional consent.

#### What are my rights if I take part in this study?

Participation in this study is voluntary. You may refuse to participate or withdraw at any time without penalty. You have the right to skip or not answer any questions you prefer not to answer.

> NYU IRB-FY2020-4194 Approved on 1-24-2025 Expires on 1-24-2026

William Tsai, Ph.D.
Assistant Professor

Applied Psychology 246 Greene St. 8<sup>th</sup> Floor New York, NY 10003 P: 212-998-4808 Will.tsai@nyu.edu

## Who can answer questions I might have about this study?

If there is anything about the study or your participation that is unclear or that you do not understand, if you have questions or wish to report a research-related problem, you may contact Dr. William Tsai at (212)998-5552, will.tsai@nyu.edu, 246 Greene St. 8th Floor, New York, NY 10003.

For questions about your rights as a research participant, you may contact the University Committee on Activities Involving Human Subjects (UCAIHS), New York University, 665 Broadway, Suite 804, New York, New York, 10012, at ask.humansubjects@nyu.edu or (212) 998-4808. Please reference the study # (IRB-FY2020-4194) when contacting the IRB (UCAIHS).

## **Agreement to Participate**

By pressing "next", you are providing your consent to participate in this study and continue with the 45-minute survey.